CLINICAL TRIAL: NCT04847960
Title: The Effect of Probiotic Lactobacillus Reuteri Prodentis Consumption on Gingival Crevicular Fluid Inflammatory Response and Metagenomic Profiles of Oral Microbiome in Orthodontic Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trisakti University (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Indonesia University (Other); BioGaia AB (Industry)
Responsible Party: Principal Investigator, Armelia Sari Widyarman, Lecturer, Head of Microbiology Department, Head of MiCORE Laboratory, Trisakti University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0191
Record Dates: First submitted 2020-12-09; First posted 2021-04-19 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects With Fixed Orthodontics
Keywords: probiotics; Lactobacillus reuterii; oral microbiome; fixed orthodontics

STUDY DESIGN:
Intervention Model Description: intervention group
Masking Description: Open label trial of BioGaia's Probiotic lozenges
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L.reuterii probiotic lozenges from BioGaia (Experimental): Subjects were willing to provide 2 samples of saliva, dental plaque and gingival fluid (gum fluid), on the first day (before consuming lozenges) and on the 14th day after the subject consumed lozenges containing L. reuteri probiotic. Probiotics are taken once a day for two weeks after breakfast and brushing their teeth.
  Interventions: Dietary Supplement: BioGaia Probiotic Lozenges

INTERVENTIONS:
Dietary Supplement: BioGaia Probiotic Lozenges — BioGaia Prodentis lozenges is a food supplement for oral health that contains patented lactic acid bacteria Limosilactobacillus reuteri (formerly known as Lactobacillus reuteri) Prodentis (a combination of strains of L. reuteri DSM 17938 and L. reuteri ATCC PTA 5289) which helps good microorganisms maintain natural balance in the mouth. This product is safe for daily use and this product can be used during pregnancy and breastfeeding. The ingredients of this product are: bulking agent (isomalt), L. reuteri DSM 17938 and L. reuteri ATCC PTA 5289, fully hydrogenated palm oil, peppermint flavoring, menthol flavoring, peppermint oil and sweetener (sucralose). One candy contains a minimum of 200 million live L. reuteri Prodentis. Net weight per candy is 800 mg. Excessive consumption can have a laxative effect due to the sweetener content in the product. This product has obtained a distribution permit in Indonesia with a BPOM number: SI194510521 with the name Probiotic Prodentis (Pro-D).

SUMMARY:
In this study, researchers will test the effectiveness of probiotic consumption against oral pathogenic bacteria and reduce the occurrence of gingival inflammation in subjects using orthodontic fixed appliances (braces).

Lactobacillus reuteri is one of the probiotic bacteria that has been identified for its health benefits. L. reuteri produces antimicrobial substances, reuterin and reutericyclin which are active against wide range of pathogenic organisms. Previously, investigator performed a pilot study on the beneficial health effect of probiotic L. reuteri containing lozenges on a few orthodontic patients and it was proven that taking this probiotic for two weeks could significantly reduce the number of pathogenic bacteria in the patients' saliva. In vitro study showed that L. reuteri has the ability to modulate the inflammatory response such as TNF alpha and interleukins. However, The ability of L. reuteri in modulating the inflammatory response viz. Interleukin 1-beta, Interleukin 6, interleukin 8, interleukin 10, TNF alpha, MMP-9 and RANKL and effect on oral metagenomic microbiome profile in patients undergoing orthodontic treatment has not been previously investigated.

Objective:

1. To evaluate the effect of consumption of L. reuteri Prodentis probiotic lozenges on the inflammatory response (inflammation) of gingival fluid.
2. To evaluate the effect of consumption of the probiotic lozenges of L. reuteri Prodentis against oral pathogens in dental plaque and saliva.

Research Benefits:

This study was conducted to observe the effectiveness of L. reuteri (ProDentis) probiotic against oral pathogenic bacteria on patients using orthodontic fixed appliance, to reduce gum inflammation and improve oral health.

DETAILED DESCRIPTION:
Rationale and background of the study

Aesthetics is a primary consideration for patients seeking orthodontic treatment. However, apart from esthetic aspects, the malalignment of teeth may also cause health concerns affecting oral function such as mastication, speech, and psychosocial problems due to impaired dentofacial aesthetics. Hence, the subjects undergoing fixed orthodontic treatment may come across several oral health related issues. The fixed orthodontic treatment is known to place the subject at risk of accumulation of heavy dental plaque which alters the symbiotic ecosystem of oral microbiome. This leads to dysbiotic oral micrbiome which harbore more pathogenic species. It has been shown pathogenic S. mutans, P. gingivalis, A. actinomycetemcomitans and C. albicans are present in orthodontic patients who do not pay enough attention to oral hygiene procedures.

S. mutans is a facultative anaerobic Gram-positive oral bacteria that has an important role in developing dental caries. P. gingivalis and A. actinomycetemcomitans are an anaerobic Gram-negative oral bacteria associated with periodontitis. Data from The National Health and Nutrition Examination Survey (NHANES III) suggest 14% orthodontic patients in the US over 20 years of age have moderate to severe periodontitis. Moreover, presence and pathogenic potential of C. albicans in periodontal pocket of these patients has been shown. C. albicans is a robust biofilm-forming organism, presenting therapeutic complication.

L. reuteri is a commensal oral probiotic bacterium, that is known to a produce antibacterial compound, reuterin. The structure of this broad-spectrum antimicrobial is related to hydroxypropionaldehyde, which formed during fermentation with glycerol. Previous studies have shown beneficial effect of reuterin against pathogenic oral bacteria. Moreover, it is safe to be used as chewing gums or yoghurts. Furthermore, previous study found that L. reuteri-containing gum was effective in reducing plaque accumulation and gingivitis in patient with moderate to severe gingivitis. Therefore, L. reuteri-containing chewing gum has considerable evidence to be used for the improvement of oral health.

Preliminary data: As a pilot study, investigators collected saliva samples from eight orthodontic patients (mean age 21 years) before and two weeks after daily probiotic consumption. A duplicate sample was collected from each subject. The results showed significant reductions in S. mutans serotype c, S. mutans serotype d, P. gingivalis, and A. actinomycetemcomitans after probiotic consumption (p<0.05).

Research gap: The ability of L. reuteri in modulating the inflammatory response viz. Interleukin 1 beta, Interleukin 6, interleukin 8, interleukin 10, TNF alpha, MMP-9 and RANKL and effect on oral metagenomic microbiome profile in patients undergoing orthodontic treatment has not been previously investigated.

Materials and methods

Lactobacillus reuteri Prodentis lozenges, along the placebos for comparison, were shipped from BioGaia, Stockholm, Sweden. Double-blinded numbering for the lozenges was done prior to shipment for the researchers to prevent bias, thus the only party that has information regarding the lozenges difference between the treatment and placebos is BioGaia. Neither the test subjects nor the researchers has the knowledge regarding the lozenges difference.

BioGaia Prodentis lozenges is a food supplement for oral health containing the patented lactic acid bacterium Limosilactobacillus reuteri (formerly known as Lactobacillus reuteri) Prodentis (a strain combination of L. reuteri DSM 17938 and L. reuteriATCC PTA 5289) that helps the good microorganisms keep a natural balance in the mouth. This product is safe for daily use and the product can be used during pregnancy and breast-feeding. Ingredients of this poduct : bulking agent (isomalt), L. reuteri DSM 17938 and L. reuteri ATCC PTA 5289, fully hydrogenated palm oil, peppermint flavor, menthol flavor, peppermint oil and sweetener (sucralose). One lozenge consists of a minimum of 200 million live L. reuteriProdentis. Net weight per lozenge, 800 mg. Excessive consumption may have laxative effects due to the content of sweeteners in the product.

Research subject:

In order to evaluate its clinical efficacy, the probiotic L. reuteri-containing lozenges will be used for the patients undergoing fixed orthodontic therapy as previously described in the pilot study. A randomized controlled trial using a parallel design with 21 subjects in the test group and 21 subjects in the control group will be conducted. The sample size calculation was performed by assuming the control group will have no change in the oral pathogens whilst the test group will have a reduction observed in the pilot study. Considering the 2-sided test with 0.05 level of significance and 80% power in detecting such differences between the two groups, 21 subjects in each group would be required.

Subjects are student volunteers or patients of Faculty of Dentistry, Trisakti University, undergoing orthodontic treatment with fixed appliance, with following inclusion criteria: age of 18-28 of either gender; undergoing orthodontic treatment with fixed appliance for the last one year; no consumption of probiotics (min. 3 months prior); no consumption of medicine such antibiotic (min 3 months prior) and PBI Score >1. The exclusion criteria are subject with systemic diseases and allergic to probiotic. Subjects were recruited by an undergoing graduate student that was part of the research team. Subject candidates that are reluctant or unwilling may directly decline the recruitment invitation wholeheartedly, therefore the volunteers that were recruited wholeheartedly agreed to become test subjects of this research. The recruited subjects will then be randomly assigned to the test.

The time for 3 samples collection was carried out approximately 15 minutes. Sampling will be carried out at the executive clinic of the Faculty of Dentistry, Trisakti University Dental Hospital. Participants will be given toothpaste and toothbrush during the study period and subjects need to brush their teeth tiwce a day. Consumption of probiotics will be done 2 weeks after orthodontics control. Samples will be collected twice: on the first day (before consuming lozenges) and the 14th day after the subject consumed lozenges containing the probiotic L. reuteri. Probiotics are taken once a day for two weeks after breakfast and brushing teeth.

Sample collection methods Prior to sample collection, it was first confirmed that every subject has undergone rapid antigen test for SARS-CoV2 detection due to the current Covid-19 pandemic (30th of September 2020), in which the result of the test must be a negative result for every patient. Negative result indicate that the subject has no past infection of SARS-CoV2. After confirmation, sample specimen from the subjects within the minimum of two-week period after orthodontics control, was collected by a dentist / medical specialist equipped with a complete set of personal protective equipment.

Saliva sample is collected using draining method. The subject is made to sit quietly while bending down the head and opened mouth to allow the saliva to drip passively from the lower lip. Saliva is collected using a sterile, pre-weighted tubes. Subjects should be in a fasting state / two hours after breakfast. Subjects should not brush their teeth for a minimum of 45 minutes prior to saliva sampling collection. After saliva collection, it is recommended to store the saliva samples at -20oC, should the analysis not be done immediately. Additionaly, it is better to aliquot and freeze samples in several tubes to avoid freeze-thaw cycles that could degradate the saliva quality.

Plaque sample is collected by swabbing all (buccal/mesial/distal/lingual/occlusal) surfaces of the individual permanent first molar using a sterile toothpick. Plaque sample was then transferred to a sterile phosphate-buffered saline (PBS). After collection, plaque sample is stored at -20oC until further analysis to be done.

Gingival crevicular fluid (GCF) sample is collected using absorbent paper strip technique. An absorbent paper strip is gently placed to a several selected site . Strip is removed after light resistance is felt, approximately after being left for 30 seconds. Multiple paper strips for one subject is pooled into several 1.5 ml microcentrifuge tube containing 100 µl PBS at 4oC. The tubes were subsequently stored at -20oC and used for further analysis.

Part I : Clinical trial to evaluate the efficacy of probiotic on gingival inflammatory response of orthodontic patients using ELISA method.

In order to evaluate its clinical efficacy, the probiotic, L. reuteri-containing lozenges will be used for the patients undergoing fixed orthodontic therapy as previously described in the pilot study. Subjects in the test group will be given two weeks of daily consumption of the probiotic lozenges administered (2x108 CFU/tablet) after breakfast and tooth brushing. Samples will be collected from all the subjects on day one and day fourteen. The gingival crevicular fluid, saliva and dental plaque samples will be collected from the recruited subjects prior to the group allocation using standard methodology as previously described [30]. The collected samples will be stored in a cooler box and placed in laboratory refrigerator at -80°C. The samples will be used to analyze the Interleukin 1-beta, Interleukin 6, interleukin 8, interleukin 10, TNF alpha, MMP-9 and RANKL level using ELISA method (BioLegend, San Diego, USA).

Part II: Clinical trial to evaluate the probiotic effect on metagenomic oral microbiome on orthodontic patients using NGS Saliva and plaque sample will be collected from each groups. Investigators will do microbiome profiling for 40 samples each sequencing run. Bacterial and fungal DNA of collected samples will be extracted using MoBio PowerSoil® DNA Isolation Kit or Qiagen QIAamp® DNA Mini Kit. Extraction method will follow the kit's manufacture protocol. Extracted DNA will be subjected to quality check using Nanodrop. Concentration of gDNA will be measured by using Qubit fluorometer. The recommended gDNA concentration from each sample is 5 ng/uL. Following quality control, V3-V4 regions of 16S and 18S rRNA gene of each sample will be amplified using PCR. During library preparation, yielded amplicons will be converted into library by using Nextera XT Index Kit (Illumina, US) accordingly to the manufacture's instruction. All resultant libraries will be evaluated by using Qubit fluorometer and will be sequenced using iSeq 100 platform (Illumina, US). Sequencing parameter will be 300 cycles with PhiX control spike-in of 5%. Visualized microbial profiling data from the sequence run can be viewed using Illumina Local Run Manager software.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 28 years old (M/F)
* Using orthodontic fixed appliance for at least 1 year
* Do not consume probiotics and antibiotics (at least 3 months before)
* No history of systemic disease

Exclusion Criteria:

* Subjects with systemic diseases
* Allergic to probiotics

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Metagenomic microbiome profile comparison between Pre- and Post-treatment described using Alpha Diversity analysis. | 8 weeks
  Using next-generation sequencing to acquire both bacterial and fungal metagenomic profile from plaque, gingival crevicular fluid, and saliva samples, whilst comparing both profile between pre-treatment and post-treatment. The data will be analysed and presented after observed operational taxonomic units (OTU), Shannon's richness, Chao's richness, and Simpson's evenness analysis has been done.
Bacterial gene expression profile from dental plaque comparison between Pre- and Post-treatment described using relative quantification of fold gene expression (2-∆∆Ct). | 16 weeks
  Using RT-PCR to acquire the gene expression of bacterial dental plaque that are acquired from both pre-treatment and post-treatment samples, therefore comparing bacterial dental plaque's gene expression between pre-treatment and post-treatment.
Proteomic profile assessed from gingival crevicular fluid and comparing its results between Pre- and Post-treatment as assessed using enzyme-linked immunosorbant assay. | 12 weeks
  Using enzyme-linked immunosorbant assay to assess inflammatory responses and comparing it between pre-treatment samples and post-treatment samples. Standard curves for each marker will also be conducted. Final protein concentrations of each marker will be generated after the sample's absorbance value detected is converted using the standard curve of each marker.
OHI status and Plaque index as assessed by the dental general practitioners. | 2 weeks
  Assessment done by dentists to analyze oral health comparisons between pre-treatment and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Armelia Sari Widyarman, Ph.D, Principal Investigator — Trisakti University; Chaminda Jayampath Seneviratne, Ph.D, Study Director — Duke-NUS Graduate Medical School; Citra Fragnantia Theodora, Ph.D, Study Chair — Indonesia University; Joko Kusnoto, Sp.Ortho, Study Chair — Trisakti University; Tri Erri Astoeti, Professor, Study Chair — Trisakti University
Locations (1):
- Trisakti University, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Saraf K, Shashikanth MC, Priy T, Sultana N, Chaitanya NC. Probiotics--do they have a role in medicine and dentistry? J Assoc Physicians India. 2010 Aug;58:488-90, 495-6. PMID 21189696
- [Background] Urbanska M, Szajewska H. The efficacy of Lactobacillus reuteri DSM 17938 in infants and children: a review of the current evidence. Eur J Pediatr. 2014 Oct;173(10):1327-37. doi: 10.1007/s00431-014-2328-0. Epub 2014 May 13. PMID 24819885
- [Background] Julien KC, Buschang PH, Campbell PM. Prevalence of white spot lesion formation during orthodontic treatment. Angle Orthod. 2013 Jul;83(4):641-7. doi: 10.2319/071712-584.1. Epub 2013 Jan 4. PMID 23289733
- [Background] Grzic R, Spalj S, Lajnert V, Glavicic S, Uhac I, Pavicic DK. Factors influencing a patient's decision to choose the type of treatment to improve dental esthetics. Vojnosanit Pregl. 2012 Nov;69(11):978-85. PMID 23311250
- [Background] Nalcaci R, Demirer S, Ozturk F, Altan BA, Sokucu O, Bostanci V. The relationship of orthodontic treatment need with periodontal status, dental caries, and sociodemographic factors. ScientificWorldJournal. 2012;2012:498012. doi: 10.1100/2012/498012. Epub 2012 Oct 23. PMID 23193381
- [Background] Pathak AK, Sharma DS. Biofilm associated microorganisms on removable oral orthodontic appliances in children in the mixed dentition. J Clin Pediatr Dent. 2013 Spring;37(3):335-9. doi: 10.17796/jcpd.37.3.92230h6256v8697t. PMID 23855182
- [Background] Özyildiz F, Uzel A, Hazar A, Güden M, Ölmez S, Aras I et al. Photocatalytic antimicrobial effect of TiO2 anatase thin-film-coated orthodontic arch wires on 3 oral pathogens. Turkish Journal of Biology. 2014;38:289-295.
- [Background] Arikan V, Kizilci E, Ozalp N, Ozcelik B. Effects of Fixed and Removable Space Maintainers on Plaque Accumulation, Periodontal Health, Candidal and Enterococcus Faecalis Carriage. Med Princ Pract. 2015;24(4):311-7. doi: 10.1159/000430787. Epub 2015 Jun 4. PMID 26044443
- [Background] Islam B, Khan SN, Khan AU. Dental caries: from infection to prevention. Med Sci Monit. 2007 Nov;13(11):RA196-203. PMID 17968308
- [Background] Marsh P, Martin M V., Lewis MAO. Oral Microbiology. 5th ed. Elsevier Ltd; 2009:78-84.
- [Background] Brigido JA, da Silveira VR, Rego RO, Nogueira NA. Serotypes of Aggregatibacter actinomycetemcomitans in relation to periodontal status and geographic origin of individuals-a review of the literature. Med Oral Patol Oral Cir Bucal. 2014 Mar 1;19(2):e184-91. doi: 10.4317/medoral.19304. PMID 24316700
- [Background] Di Benedetto A, Gigante I, Colucci S, Grano M. Periodontal disease: linking the primary inflammation to bone loss. Clin Dev Immunol. 2013;2013:503754. doi: 10.1155/2013/503754. Epub 2013 May 23. PMID 23762091
- [Background] Karkhanechi M, Chow D, Sipkin J, Sherman D, Boylan RJ, Norman RG, Craig RG, Cisneros GJ. Periodontal status of adult patients treated with fixed buccal appliances and removable aligners over one year of active orthodontic therapy. Angle Orthod. 2013 Jan;83(1):146-51. doi: 10.2319/031212-217.1. Epub 2012 Jun 22. PMID 22725616
- [Background] Canabarro A, Valle C, Farias MR, Santos FB, Lazera M, Wanke B. Association of subgingival colonization of Candida albicans and other yeasts with severity of chronic periodontitis. J Periodontal Res. 2013 Aug;48(4):428-32. doi: 10.1111/jre.12022. Epub 2012 Nov 8. PMID 23137301
- [Background] Cruz MR, Graham CE, Gagliano BC, Lorenz MC, Garsin DA. Enterococcus faecalis inhibits hyphal morphogenesis and virulence of Candida albicans. Infect Immun. 2013 Jan;81(1):189-200. doi: 10.1128/IAI.00914-12. Epub 2012 Oct 31. PMID 23115035
- [Background] Jones SE, Versalovic J. Probiotic Lactobacillus reuteri biofilms produce antimicrobial and anti-inflammatory factors. BMC Microbiol. 2009 Feb 11;9:35. doi: 10.1186/1471-2180-9-35. PMID 19210794
- [Background] Cleusix V, Lacroix C, Vollenweider S, Le Blay G. Glycerol induces reuterin production and decreases Escherichia coli population in an in vitro model of colonic fermentation with immobilized human feces. FEMS Microbiol Ecol. 2008 Jan;63(1):56-64. doi: 10.1111/j.1574-6941.2007.00412.x. Epub 2007 Nov 20. PMID 18028400
- [Background] Vollenweider S, Lacroix C. 3-hydroxypropionaldehyde: applications and perspectives of biotechnological production. Appl Microbiol Biotechnol. 2004 Mar;64(1):16-27. doi: 10.1007/s00253-003-1497-y. Epub 2003 Dec 11. PMID 14669058
- [Background] Caglar E, Cildir SK, Ergeneli S, Sandalli N, Twetman S. Salivary mutans streptococci and lactobacilli levels after ingestion of the probiotic bacterium Lactobacillus reuteri ATCC 55730 by straws or tablets. Acta Odontol Scand. 2006 Oct;64(5):314-8. doi: 10.1080/00016350600801709. PMID 16945898
- [Background] Nikawa H, Makihira S, Fukushima H, Nishimura H, Ozaki Y, Ishida K, Darmawan S, Hamada T, Hara K, Matsumoto A, Takemoto T, Aimi R. Lactobacillus reuteri in bovine milk fermented decreases the oral carriage of mutans streptococci. Int J Food Microbiol. 2004 Sep 1;95(2):219-23. doi: 10.1016/j.ijfoodmicro.2004.03.006. PMID 15282133
- [Background] Iniesta M, Herrera D, Montero E, Zurbriggen M, Matos AR, Marin MJ, Sanchez-Beltran MC, Llama-Palacio A, Sanz M. Probiotic effects of orally administered Lactobacillus reuteri-containing tablets on the subgingival and salivary microbiota in patients with gingivitis. A randomized clinical trial. J Clin Periodontol. 2012 Aug;39(8):736-44. doi: 10.1111/j.1600-051X.2012.01914.x. Epub 2012 Jun 13. PMID 22694350
- [Background] Teughels W, Newman MG, Coucke W, Haffajee AD, Van Der Mei HC, Haake SK, Schepers E, Cassiman JJ, Van Eldere J, van Steenberghe D, Quirynen M. Guiding periodontal pocket recolonization: a proof of concept. J Dent Res. 2007 Nov;86(11):1078-82. doi: 10.1177/154405910708601111. PMID 17959900
- [Background] Shimauchi H, Mayanagi G, Nakaya S, Minamibuchi M, Ito Y, Yamaki K, Hirata H. Improvement of periodontal condition by probiotics with Lactobacillus salivarius WB21: a randomized, double-blind, placebo-controlled study. J Clin Periodontol. 2008 Oct;35(10):897-905. doi: 10.1111/j.1600-051X.2008.01306.x. Epub 2008 Aug 24. PMID 18727656
- [Background] Morita H, Toh H, Fukuda S, Horikawa H, Oshima K, Suzuki T, Murakami M, Hisamatsu S, Kato Y, Takizawa T, Fukuoka H, Yoshimura T, Itoh K, O'Sullivan DJ, McKay LL, Ohno H, Kikuchi J, Masaoka T, Hattori M. Comparative genome analysis of Lactobacillus reuteri and Lactobacillus fermentum reveal a genomic island for reuterin and cobalamin production. DNA Res. 2008 Jun 30;15(3):151-61. doi: 10.1093/dnares/dsn009. Epub 2008 May 16. PMID 18487258
- [Background] Krasse P, Carlsson B, Dahl C, Paulsson A, Nilsson A, Sinkiewicz G. Decreased gum bleeding and reduced gingivitis by the probiotic Lactobacillus reuteri. Swed Dent J. 2006;30(2):55-60. PMID 16878680
- [Background] Twetman S, Derawi B, Keller M, Ekstrand K, Yucel-Lindberg T, Stecksen-Blicks C. Short-term effect of chewing gums containing probiotic Lactobacillus reuteri on the levels of inflammatory mediators in gingival crevicular fluid. Acta Odontol Scand. 2009;67(1):19-24. doi: 10.1080/00016350802516170. PMID 18985460

DOCUMENTS (2):
  • Study Protocol (2021-01-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT04847960/Prot_000.pdf
  • Informed Consent Form (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT04847960/ICF_001.pdf